CLINICAL TRIAL: NCT03483207
Title: Acute Mesenteric Venous Thrombosis.. in Assiut University Hospital Management Controversies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dr. Hamada, Resident at General surgery department, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HF2018
Record Dates: First submitted 2018-01-20; First posted 2018-03-30 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-01

CONDITIONS: Mesenteric Vein Thrombosis
MeSH Terms: conditions — Mesenteric Ischemia | interventions — Warfarin; Heparin

STUDY DESIGN:
Intervention Model Description: Diagnosis of acute MVT will be based on clinical presentation &positive CT scan.(9) .patients with confirmed diagnosis of acute MVT on CT scan but having no signs of peritonitis or established CT signs of gangrene will be treated conservatively .(11)In addition to usual care ,intravenous heparin will be started and the dose is adjusted to maintain APTT levels at 2-2.5 times the normal. (12) followed by oral anticoagulation (warfarin) for 6 months or for life in the presence of coagulation abnormality. All patients will be critically monitored for the progress of response of therapy , failure to improve or worsening in condition,will be an urgent indication for surgical intervention with resection of the infarcted bowel segment .If there is suspicion about the viability of remaining bowel intraoperative or later on based on clinical evidences,then" second look" laparotomy will be perfomed .The mortality and all complications associated with surgery will be recorded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MVT with anticoagulation therapy(heparin &warfarin) (Experimental): patients with confirmed diagnosis of acute MVT on CT scan but having no signs of peritonitis or established CT signs of gangrene will be treated conservatively with anticoagulation(heparin &warfarin) while other cases will be for surgical management and not included in the study.
  Interventions: Drug: Warfarin; Procedure: MVT with failure of anticoagulation therapy; Drug: Heparin
- MVT with failure of anticoagulation therapy(heparin &warfarin) (Experimental): patients who underwent conservative therapy with anticoagulation (heparin &warfarin) but showed no improvement .
  Interventions: Drug: Warfarin; Procedure: MVT with failure of anticoagulation therapy; Drug: Heparin

INTERVENTIONS:
Drug: Warfarin — Patients with confirmed diagnosis of acute MVT but having no signs of bowel infarction will be treated conservatively with anticoagulation (heparin &warfarin) In addition to usual care intravenous low molecular weight heparin will be started (IV bolus of 5000 IU followed by 1000 IU/hour with infusion pump) and the dose is adjusted to maintain APTT levels at 2-2.5 times the normal. followed by oral anticoagulation (warfarin) for 6 months or for life in the presence of coagulation abnormality. patients will be critically monitored for the progress of response of therapy .
Procedure: MVT with failure of anticoagulation therapy — patients managed conservatively with anticoagulation will be monitored for the progress of response of therapy , failure to improve or worsening in condition,will be an urgent indication for surgical intervention with resection of the infarcted bowel segment .If there is suspicion about the viability of remaining bowel intraoperative or later on based on clinical evidences,then" second look" laparotomy will be performed .The mortality and all complications associated with surgery will be recorded.
Drug: Heparin — Patients with confirmed diagnosis of acute MVT but having no signs of bowel infarction will be treated conservatively with anticoagulation (heparin &warfarin) In addition to usual care intravenous low molecular weight heparin will be started (IV bolus of 5000 IU followed by 1000 IU/hour with infusion pump) and the dose is adjusted to maintain APTT levels at 2-2.5 times the normal. followed by oral anticoagulation (warfarin) for 6 months or for life in the presence of coagulation abnormality. patients will be critically monitored for the progress of response of therapy .

SUMMARY:
Initial treatment in the management of acute mesenteric vein thrombosis (MVT) is controversial. Some authors have proposed a surgical approach, whereas others have advocated medical therapy (anticoagulation). In this study, the investigators analyzed and compared the results obtained with surgical and medical treatment to determine the best initial management for this disease.

DETAILED DESCRIPTION:
Mesenteric venous thrombosis (MVT) is increasingly recognized as a cause of mesenteric ischemia. it must be distinguished from arterial and non occlusive types of ischemia, it accounts for 5% to 15% of all cases of mesenteric ischemia. Patients may have evocative signs,such as abdominal pain that is out of proportion to physical signs, nausea, or vomiting. However, a clinical diagnosis is often difficult because abdominal symptoms are non specific and high index of suspicion is often required for diagnosis.(1) Primary MVT accounted for 25% to 55% of cases in early studies, but recent reports show decline in primary MVT because of improvements in the diagnosis of hypercoagulable states.(2) Advances in new imaging techniques also have enabled early recognition of this disease without or before laparotomy.(3-5 ) Fortunately , there is no consensus about the initial management of MVT; Some authors have proposed an aggressive surgical approach (6) while others have advocated an initial conservative management with anticoagulation and close monitoring . ( 7) similarly,issue of second look laparotomy,mandatory or selective is yet not resolved.

The present study is prompted to analyze our experience in an effort to resolve these controversies and the results obtained will be assessed to determine the best management strategy for this uncommon disease.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients admitted in the department of surgery in Assiut University diagnosed to have mesenteric venous occlusion not presented by signs of peritonitis or confirmed radiological signs of bowel infarction.

Exclusion Criteria:

1-Patients diagnosed to have mesenteric venous occlusion but with signs of peritonitis or confirmed radiological signs of bowel infarction on admission.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Anticoagulation therapy (heparin &warfarin) in MVO | within 3-6 months of starting treatment.
  patients with confirmed diagnosis of acute MVT on CT scan will be treated conservatively In addition to usual care such as fluid and electrolyte balance, antibiotic coverage and nasogastric intubation ,intravenous heparin will be started and the dose is adjusted to maintain APTT levels at 2-2.5 times the normal. followed by oral anticoagulation (warfarin) for 6 months or for life in the presence of coagulation abnormality. All patients will be critically followed up(Clinically.. Radiologically ) for the progress of response of therapy , failure to improve or worsening in condition( appearance of signs of peritonitis such as guarding, rigidity and fever...or radiological signs of bowel infarction) will be assessed .
  Factors that may affect the response such as ( age, duration from onset of the disease till starting therapy,underlying diseases,.. )also complications (hemorrhage, failure ,..)will be assessed

SECONDARY OUTCOMES:
Recurrence rate | within six months of starting treatment.
  number of recurrent cases post conservative therapy .
Mortality rate | within one year of starting treatment.
  number of deaths as a complication of conservative therapy or surgery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grendell JH, Ockner RK. Mesenteric venous thrombosis. Gastroenterology. 1982 Feb;82(2):358-72. No abstract available. PMID 7033036
- [Background] Zhang J, Duan ZQ, Song QB, Luo YW, Xin SJ, Zhang Q. Acute mesenteric venous thrombosis: a better outcome achieved through improved imaging techniques and a changed policy of clinical management. Eur J Vasc Endovasc Surg. 2004 Sep;28(3):329-34. doi: 10.1016/j.ejvs.2004.06.001. PMID 15288639
- [Background] Harnik IG, Brandt LJ. Mesenteric venous thrombosis. Vasc Med. 2010 Oct;15(5):407-18. doi: 10.1177/1358863X10379673. PMID 20926500
- [Background] Harward TR, Green D, Bergan JJ, Rizzo RJ, Yao JS. Mesenteric venous thrombosis. J Vasc Surg. 1989 Feb;9(2):328-33. PMID 2918628
- [Background] Prout WG. The significance of rebound tenderness in the acute abdomen. Br J Surg. 1970 Jul;57(7):508-10. doi: 10.1002/bjs.1800570706. No abstract available. PMID 5427470
- [Background] Rhee RY, Gloviczki P, Mendonca CT, Petterson TM, Serry RD, Sarr MG, Johnson CM, Bower TC, Hallett JW Jr, Cherry KJ Jr. Mesenteric venous thrombosis: still a lethal disease in the 1990s. J Vasc Surg. 1994 Nov;20(5):688-97. doi: 10.1016/s0741-5214(94)70155-5. PMID 7966803
- [Background] Kumar S, Kamath PS. Acute superior mesenteric venous thrombosis: one disease or two? Am J Gastroenterol. 2003 Jun;98(6):1299-304. doi: 10.1111/j.1572-0241.2003.07338.x. PMID 12818273
- [Background] Pabinger I, Schneider B. Thrombotic risk in hereditary antithrombin III, protein C, or protein S deficiency. A cooperative, retrospective study. Gesellschaft fur Thrombose- und Hamostaseforschung (GTH) Study Group on Natural Inhibitors. Arterioscler Thromb Vasc Biol. 1996 Jun;16(6):742-8. doi: 10.1161/01.atv.16.6.742. PMID 8640401
- [Background] Brunaud L, Antunes L, Collinet-Adler S, Marchal F, Ayav A, Bresler L, Boissel P. Acute mesenteric venous thrombosis: case for nonoperative management. J Vasc Surg. 2001 Oct;34(4):673-9. doi: 10.1067/mva.2001.117331. PMID 11668323